CLINICAL TRIAL: NCT05598749
Title: Evaluation of the Immunomodulation Effect of ESIT12, a Poplar-type Propolis Dry Extract and Its Efficacy in Subjects At Risk of Contracting Upper Respiratory Tract Infections (URTIs)
Brief Title: Poplar-type Propolis Dry Extract ESIT12 : Immunomodulation Efficacy Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fytexia (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: ESIT12IES
Record Dates: First submitted 2022-10-25; First posted 2022-10-28 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-09

CONDITIONS: Upper Respiratory Tract Infection (URTI)
MeSH Terms: conditions — Respiratory Tract Infections | interventions — calcium D-pantothenate, L-cysteine drug combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo
- Verum (Experimental)
  Interventions: Dietary Supplement: Verum

INTERVENTIONS:
Dietary Supplement: Placebo — Arabic gum, sucrose and silicon dioxide mix
  Arms: Placebo
Dietary Supplement: Verum — Propolis dry extract ESIT12 and carriers (arabic gum, sucrose and silicon dioxide mix)
  Arms: Verum

SUMMARY:
The aim of the present investigation is to evaluate the immunomodulation effect of ESIT12, a poplar-type propolis dry extract standardized in polyphenols, and its efficacy in subjects at risk of contracting upper respiratory tract infections (URTIs), during a 12-week supplementation period plus 4-week follow-up.

The number of onset of upper respiratory tract infections, the symptoms severity and lasting and interferences with well-being will be assessed with WURSS-24 questionnaire. The quality of life will be assessed with the SF-36 questionnaire and a testimonial. Blood immune markers will also be assessed. Finally, long lasting benefits will additionally be evaluated 4 weeks after end of the supplementation period. The design of the study is double-blind, randomized, parallel and placebo controlled.

ELIGIBILITY:
Inclusion Criteria:

* inactive or minimally active according to the IPAQ short form questionnaire
* BMI 18,5-29,9

Exclusion Criteria:

* Pregnant women, breastfeeding women, women positive at Beta-HCG serology test and who hope to become pregnant
* Allergy to beehive products and known allergy (general)
* Cystic fibrosis
* Congenital or acquired immunodeficiency syndrome and disease
* History of asthma (within prior 24 months) or chronic respiratory disease
* Subjects who underwent medical treatment for COVID-19 within last 3 months
* History of immune system disorder or auto-immune disorder
* History of treated diabetes or treated hypertension
* Evidence or history of hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, neurologic diseases, and malignancies
* Cancers
* Those considered unsuitable for the participation by the physician
* No vaccination within 12 weeks prior to enrolling in the study
* No antibiotics within 12 weeks prior to enrolling in the study
* No anti-inflammatory drugs within 4 weeks prior to enrolling in the study
* No steroids within 12 weeks prior to enrolling in the study
* No immunological drugs within 4 weeks prior to enrolling in the study
* No food/dietary supplements within 4 weeks prior to enrolling in the study
* No current or recent participation in another clinical trial (within 30 days prior to screening)

Ages: 25 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 309 (Actual)
Dates: Start 2022-12-05 (Actual); Primary Completion 2024-07-03 (Actual); Study Completion 2024-07-03 (Actual)

PRIMARY OUTCOMES:
Supplementation Efficacy on URTI incidence | 12 weeks
  The incidence of URTI developped in Verum compare to Placebo measured with the WURSS-24 symptoms questionnaire
Supplementation Efficacy on number of URTI incidence | 12 weeks
  The number of URTI incidence per person in Verum compare to Placebo measured with the WURSS-24 symptoms questionnaire

SECONDARY OUTCOMES:
Supplementation Efficacy on URTI symptoms | 12 weeks
  The comparison of symptoms score (domain 2) between placebo and verum as measured with WURSS-24 questionnaire
Supplementation Efficacy on impact of URTI on quality of life | 12 weeks
  The comparison of cold-specific functional impairments (domain 3) between placebo and verum as measured with WURSS-24 questionnaire
Supplementation Efficacy on URTI severity | 12 weeks
  The comparison of global cold severity (domain 4) between placebo and verum as measured with WURSS-24 questionnaire
Supplementation Efficacy on immunomodulation | 12 weeks
  Assessment of immunological vigor (SIV) as monitored by 4 PBMC panels Panel 1 : global activation Panel 2 : Tcells focus Panel 3 : B cells focus Panel : Neutrophils / monocytes focus

CONTACTS AND LOCATIONS:
Overall Officials: Pedro Alcaraz, Principal Investigator — UCAM (Universidad Catolica San Antonio de Murcia)
Locations (1):
- UCAM (Universidad Catolica San Antonio de Murcia), Murcia, Spain

IPD SHARING:
Plan to Share IPD: No